CLINICAL TRIAL: NCT06839001
Title: Cryoablation Versus Breast Surgery in the Local Treatment of Early-Stage Breast Cancer - Six Trial
Brief Title: CRYoablation for Small Tumors As Local Treatment - SIX Trial
Acronym: CRYSTAL - SIX
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Responsible Party: Principal Investigator, Vanessa Monteiro Sanvido, Vanessa Monteiro Sanvido, Hospital do Coracao
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7.241.846
Record Dates: First submitted 2025-02-16; First posted 2025-02-21 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Breast Neoplasm
Keywords: Breast Cancer; Minimally Invasive Surgical Procedures; Cryoablation; Locoregional Recurrence; Cost-Minimization Analysis
MeSH Terms: conditions — Breast Neoplasms | interventions — Cryosurgery; Mastectomy, Segmental; Mastectomy

STUDY DESIGN:
Intervention Model Description: The initial 750 participants will be randomized in a 1:1 manner to either cryoablation or breast surgery. This is a Phase 3 randomized trial evaluating the efficacy and safety of cryoablation compared to breast surgery for early-stage breast cancer. Although the intervention does not involve drugs or biologics, it meets the criteria of a Phase 3 trial as a confirmatory study of an interventional procedure.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cryoablation (Experimental): Patients will be treated with cryoablation using a Cryoprobe under real-time ultrasound guidance and local anesthesia. The cryoablation procedure consists of a freezing phase followed by passive thawing, ending with a second freezing cycle. It is recommended to use 6 minutes of freezing and 4 minutes of thawing with Cryocare, and 10 minutes of freezing and 10 minutes of thawing with ProSense IceCure®. The freeze-thaw-freeze times may be adjusted at the physician's discretion depending on tumor size. Patients will be treated with cryoablation (Day 1) using a single Cryoprobe, followed by adjuvant treatment. In cases where radiotherapy is indicated, the preferred regimen will be the 5-fraction schedule. If the 5-fraction regimen is not feasible, the radiation oncologist will be allowed to adjust the fractionation as needed. Patients assigned to the cryoablation group will not undergo axillary surgery, as axillary surgery will be omitted.
- Breast Surgery (Lumpectomy or Mastectomy) (Active Comparator): Surgery will be performed under general anesthesia according to standard operative procedures at the hospital of origin. Surgery may be performed as either a lumpectomy or a mastectomy, along with a sentinel lymph node biopsy. After surgery, patients will undergo adjuvant treatment as indicated. If radiotherapy is required, the preferred regimen will be the 5-fraction schedule. If the 5-fraction regimen is not feasible, the radiation oncologist will be allowed to adjust the fractionation as needed.
  Interventions: Procedure: Breast Surgery (Lumpectomy or Mastectomy)

INTERVENTIONS:
Procedure: cryoablation — Two devices can be used to perform cryoablation: Cryocare® and ProSense IceCure®:
  * Cryocare® - This procedure utilizes two types of gases: argon gas for freezing and helium gas for thawing.
  * ProSense IceCure® - This procedure uses extremely low temperatures generated by liquid nitrogen (LN2) to freeze and destroy the target tissue, without the need for an additional gas.
Procedure: Breast Surgery (Lumpectomy or Mastectomy) — Surgery can be performed as lumpectomy or mastectomy and axillary surgery, preferably sentinel lymph node biopsy.
  Arms: Breast Surgery (Lumpectomy or Mastectomy)

SUMMARY:
To demonstrate the non-inferiority of cryoablation compared to breast surgery for the local treatment of early-stage breast cancer and to conduct a cost-minimization analysis comparing direct costs between treatments.

DETAILED DESCRIPTION:
This study compares cryoablation with breast surgery for the treatment of early-stage breast cancer (T1N0M0), evaluating locoregional recurrence, cost-minimization, and disease-free survival.

The primary objective is to demonstrate the non-inferiority of cryoablation compared to breast surgery for local treatment of early-stage breast cancer over five years, as well as to perform a cost-minimization analysis to compare the direct costs of both treatments over one year.

The secondary objectives include assessing locoregional recurrence at one year, evaluating disease-free survival and overall survival over five years, analyzing circulating tumor cells (CTCs) as prognostic factors and for monitoring cryoablation at baseline (study inclusion), six months, and twelve months, measuring patient satisfaction one year after randomization using the Breast-Q questionnaire, and assessing quality of life using the EQ-5D questionnaire.

Cryoablation is a nonsurgical, minimally invasive technique that destroys tumor tissue through cyclic freezing and thawing using cryoprobes. This process induces cellular death without requiring hospitalization, allowing for faster recovery.

Additionally, the study incorporates a de-escalated and personalized approach to breast cancer treatment by omitting sentinel lymph node biopsy, integrating ultrahypofractionated radiotherapy, and utilizing liquid biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Unifocal primary invasive breast carcinoma
* Tumor size ≤ 2.0 cm (T1)
* Complete pathological report (including results for ER, PR, HER2, Ki-67, and FISH report for the ERBB2 gene, if necessary)
* Lesion visible on ultrasound
* Surgical treatment would be the first option, regardless of immunohistochemistry results

Exclusion Criteria:

* Multifocal or multicentric invasive breast carcinoma
* Ductal carcinoma in situ
* Breast cancer with skin involvement
* Clinically positive axilla (N1, N2 or N3)
* Distance from lesion and skin less than 5 mm
* Prior neoadjuvant systemic therapy for breast cancer
* Distant metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Locoregional recurrence (LRR) | 5 years
  LRR was defined as recurrence in the ipsilateral breast or chest wall, as well as in the ipsilateral axillary, supraclavicular/infraclavicular region, or internal mammary lymph nodes detected during follow-up, regardless of whether distant metastasis occurred before, after, or simultaneously.
Cost-minimization | 1 year
  A cost-minimization analysis is an economic technique used to compare the costs of different interventions or treatments that produce equivalent outcomes in terms of efficacy and clinical effects. In other words, this analysis is applied when treatments are assumed to have the same clinical effectiveness, and the goal is to determine which one has the lowest cost. It is a type of cost-effectiveness analysis that compares only the costs of two or more technologies, as the health effects resulting from the compared technologies are considered similar. Clinical outcomes will not be taken into account. We will calculate the costs by collecting data on both direct and indirect expenses associated with the treatments. Direct costs will include procedure-related expenses such as equipment, supplies, medical fees, associated tests and consultations, hospitalization costs if applicable, and medication use. Indirect costs, if a societal perspective is considered, will include factors such as ti

SECONDARY OUTCOMES:
Locoregional recurrence (LRR) | 1 year
  LRR was defined as recurrence in the ipsilateral breast or chest wall, as well as in the ipsilateral axillary, supraclavicular/infraclavicular region, or internal mammary lymph nodes detected during follow-up, regardless of whether distant metastasis occurred before, after, or simultaneously.
Disease-free survival (DFS) | 5 years
  DFS is defined as the time from procedure to time of ipsilateral recurrence, contralateral recurrence, regional recurrence or distant metastasis, or date of last follow-up if none of the recurrence events occur.
Overall Survival (OS) | 5 years
  OS is defined as the time from the date of first dose to the date of death due to any cause.
Circulating tumor cells (CTCs) | 1 year
  CTCs are tumor cells that have sloughed off the primary tumor and extravasate into and circulate in the blood. Blood samples will be collected from participants included in the study at the time of the procedure, at 6 months, and at 1 year. A total of 10 mL of blood will be drawn via peripheral venipuncture into EDTA tubes (BD Vacutainer®), which will be maintained under homogenization for up to 6 hours at room temperature until filtration is performed (ISET®; Rarecells Diagnostics, Paris, France). CTCs will be identified through cytopathological analysis. After filtration, membranes washed with PBS and air-dried will be stored at -20°C until analysis. Blood samples for CTC research will preferably be sent within 48 hours and no later than 72 hours to the coordinating center.
Patient satisfaction | 1 month
  Patient satisfaction will be assessed using the Breast-Q questionnaire, a validated tool designed to measure patient-reported outcomes related to breast surgery and treatment.
EQ-5D questionnaire | 1 year
  Quality of life will be assessed using the EQ-5D questionnaire. The EQ-VAS (Visual Analogue Scale) thermometer is a component of the EQ-5D, a standardized instrument for measuring health-related quality of life. In the EQ-VAS, patients evaluate their own health status at a given moment using a numerical scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Monteiro Sanvido, PhD, Principal Investigator — Research Institute - Hospital do Coracao; Afonso Celso Pinto Nazário, PhD, Principal Investigator — Research Institute - Hospital do Coracao; Alexandre Biasi Cavalcante, PhD, Study Director — Research Institute - Hospital do Coracao
Locations (1):
- Research Institute - Hospital do Coracao, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No